CLINICAL TRIAL: NCT05213910
Title: Study of a Management Strategy of Functional Bowel Disordes Related to Irritable Bowel Syndrome (IBS) With a Mixture of 8 Microbiotic Strains
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: PiLeJe (Industry)
Responsible Party: Sponsor
Organization: Larena SAS (Industry)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Pil-LACCB-017
Record Dates: First submitted 2021-12-13; First posted 2022-01-28 (Actual); Last update posted 2022-04-06 (Actual); Status verified 2021-12

CONDITIONS: Irritable Bowel Syndrome
MeSH Terms: conditions — Irritable Bowel Syndrome

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Patients using the product (Experimental)
  Interventions: Dietary Supplement: Lactichoc; Other: Stool sampling

INTERVENTIONS:
Dietary Supplement: Lactichoc — dosage form: mix of 8 strains containing 1.2x10^11 CFU frequency, and duration: 2 capsules/day during 10 days
Other: Stool sampling — 3 stool samples are taken during the study (D0, D10 and D30)

SUMMARY:
The aim of this study is to determine the impact of a 10-day treatment with Lactichoc® on irritable bowel syndrome.

ELIGIBILITY:
Inclusion Criteria:

* Having IBS symptomatology meeting the Rome IV criteria;
* Having a IBS-SSS score ≥150 ;
* In a state of general and mental health compatible with participation in the study ;
* Agreeing to maintain their lifestyle during the study (same dietary and physical activity habits) ;
* Willing to take stool samples;
* Able and willing to participate in the research by complying with the protocol procedures, especially regarding the consumption of the study product;
* Having electronic tools (computer, tablet...) and an internet connection, allowing him/her to fill out the self-questionnaires of the study online;
* Affiliated to a social security system.

Exclusion Criteria:

* Have a history of hypersensitivity to any of the ingredients of the study product;
* Under antibiotic treatment, or having stopped it for less than 14 days;
* Under dietary supplementation (prebiotics or probiotics) or having stopped it for less than one month;
* Having initiated or modified a background treatment for a comorbidity for less than one month, or planning to initiate it during the study, or planning to interrupt it during the study;
* Having a lifestyle incompatible with the study as determined by the investigator;
* Women who are pregnant or breastfeeding or who intend to become pregnant within the next 2 months;
* Planning to travel extensively during the study period or unable to be contacted in case of emergency;
* Psychologically or linguistically unable to understand and sign the informed consent;
* Participating in another clinical trial or on an exclusion period from a previous clinical trial;
* Under legal protection (guardianship, curatorship) or deprived of their rights following an administrative or judicial decision.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 189 (Actual)
Dates: Start 2018-09-04 (Actual); Primary Completion 2021-11-15 (Actual); Study Completion 2021-11-15 (Actual)

PRIMARY OUTCOMES:
Evolution of the severity of functional bowel disorders | 10 days
  The severity of functional bowel syndrome is evaluated by Irritable Bowel Syndrome Severity Scoring System (IBS-SSS)

SECONDARY OUTCOMES:
Evolution of the severity of functional bowel disorders | Between V2 (Day10) and Day30 (20 days)
  The severity of functional bowel syndrome is evaluated by Irritable Bowel Syndrome Severity Scoring System (IBS-SSS)
Description of the symptomatology | V1(Day0), V2 (Day10) and Day30
  - 10-day average stool consistency according to the Bristol Stool Scale;
Description of the symptomatology | V1(Day0), V2 (Day10) and Day30
  - 10-day average daily stool frequency;
Description of the symptomatology | V1(Day0), V2 (Day10) and Day30
  - 10-day average abdominal pain score (Irritable Bowel Syndrome Severity Scoring System (IBS-SSS) item 1b);
Description of the symptomatology | V1(Day0), V2 (Day10) and Day30
  - 10-day global self-assessment of the impact of IBS symptoms (Irritable Bowel Syndrome Severity Scoring System (IBS-SSS) item 4)
Description of quality of life | V1(Day0), V2 (Day10) and Day30
  Evaluated by the GIQLI (Gastrointestinal Quality of Life Index)
Description of the anxiety-depressive disorders | V2 (Day10)
  Evaluated by the Hospital Anxiety and Depression (HAD) scale
Safety (tolerance to treatment) | V2 (Day10)
  Calculated with adverse events that may be observed during study period (descriptif results)
Treatment compliance | V2 (Day10)
  By counting treatments returned at the V2 visit
Global clinical evaluation | V2 (Day10)
  Evaluated by the investigator (V2) by a questionnaire
Global clinical evaluation | V2 (Day10) and Day30
  Evaluated by the patient (V2 and D30) by a questionnaire
Evaluation of the satisfaction concerning the product by a questionnaire | Day30
  Evaluated by the patient

OTHER OUTCOMES:
Evolution of the stool microbiota composition | Between V1 (Day0) and V2 (Day10), then V2 (Day10) and Day30
  Metagenomic analysis

CONTACTS AND LOCATIONS:
Overall Officials: Dominique DELSART, Principal Investigator
Locations (1):
- General practitioners or gastroenterologists consulting in french private offices, Paris, France

IPD SHARING:
Plan to Share IPD: No